CLINICAL TRIAL: NCT07076836
Title: Zusanli (ST36) Electroacupuncture Treatment for Neoadjuvant Immunotherapy in Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xuelei Ma MD, Deputy Director (Medical) of the Department of Biotherapy, Cancer Center, West China Hospital, Sichuan University; Associate Director of the Stem Cell Research and Translational Research Laboratory; PhD Supervisor; Professor/Researcher, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Approval No. 2030 (2023)
Record Dates: First submitted 2025-06-26; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer (NSCLC); Small Cell Lung Cancer ( SCLC ); Immune Checkpoint Blockade; Electroacupuncture
Keywords: lung cancer (NSCLC); small cell lung cancer (SCLC); immune checkpoint blockade; electroacupuncture
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Acupuncture Therapy; Drug Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient did not know in advance whether the use of electroacupuncture or false acupuncture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental)
  Interventions: Device: Acupuncture
- Sham electroacupuncture group (Experimental)
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: Acupuncture — The electroacupuncture parameters were set as follows: frequency at 10 Hz, current intensity at 0.5 mA, pulse width at 50 μs, and each session lasted 30 minutes. On the first day of chemotherapy, electroacupuncture was administered 1-2 hours prior to chemotherapy initiation. From Day 2 to the final day of chemotherapy, electroacupuncture sessions were conducted daily between 2:00 PM and 4:00 PM.
  Other Names: ICIs; chemotherapy
  Arms: Electroacupuncture group
Device: sham acupuncture — The sham electroacupuncture group referenced the same acupoints as the electroacupuncture group, but the false acupoint shallow needling method and false electrode method are used, and the treatment time and course are the same as the electroacupuncture group.
  Other Names: ICIs
  Arms: Sham electroacupuncture group

SUMMARY:
This study aims to investigate the potential synergistic effects of acupuncture combined with immune checkpoint inhibitors in cancer therapy. Over the past decade, significant progress in cancer immunotherapy has been driven by breakthroughs in understanding immune checkpoint molecules; however, monotherapy with immune checkpoint inhibitors still faces challenges due to low response rates. As a traditional Chinese medical intervention, acupuncture modulates neuro-immune pathways to achieve remote regulation of organ functions, with particular anti-tumor potential observed at the Zusanli (ST36) acupoint-a site located 2 cm below the knee that can be stimulated via electroacupuncture (EA) to improve gastrointestinal function and alleviate inflammation. Preclinical evidence demonstrates that EA suppresses tumor growth in breast cancer models, reduces levels of pro-inflammatory cytokines such as IL-1β and TNF-α, enhances anti-tumor activity of CD8+ T cells and NK cells, and decreases accumulation of immunosuppressive myeloid-derived suppressor cells (MDSCs). Animal studies show that ST36 EA increases key immunomodulatory factors like serum IFN-γ, IL-2, and IL-17, thereby potentiating the efficacy of anti-tumor drugs. Guided by the traditional TCM principle of "reinforcing healthy qi to consolidate the body's resistance," modern clinical applications of EA combined with specific acupoint regimens (e.g., ST36, Sanyinjiao) have effectively alleviated cancer-related pain, chemotherapy-induced side effects, and fatigue. This study will evaluate the safety and immunosensitization effects of ST36 EA combined with PD-1 inhibitors in non-small cell lung cancer patients, employing 1 mA electroacupuncture for 3 consecutive days to activate immune responses. By leveraging acupuncture-induced immune remodeling, this approach aims to provide a novel integrative medicine strategy to overcome resistance to immunotherapy.

DETAILED DESCRIPTION:
This study aims to investigate the potential synergistic effects of acupuncture combined with immune checkpoint inhibitors in cancer therapy. Over the past decade, significant progress in cancer immunotherapy has been driven by breakthroughs in understanding immune checkpoint molecules; however, monotherapy with immune checkpoint inhibitors still faces challenges due to low response rates. As a traditional Chinese medical intervention, acupuncture modulates neuro-immune pathways to achieve remote regulation of organ functions, with particular anti-tumor potential observed at the Zusanli (ST36) acupoint-a site located 2 cm below the knee that can be stimulated via electroacupuncture (EA) to improve gastrointestinal function and alleviate inflammation. Preclinical evidence demonstrates that EA suppresses tumor growth in breast cancer models, reduces levels of pro-inflammatory cytokines such as IL-1β and TNF-α, enhances anti-tumor activity of CD8+ T cells and NK cells, and decreases accumulation of immunosuppressive myeloid-derived suppressor cells (MDSCs). Animal studies show that ST36 EA increases key immunomodulatory factors like serum IFN-γ, IL-2, and IL-17, thereby potentiating the efficacy of anti-tumor drugs. Guided by the traditional TCM principle of "reinforcing healthy qi to consolidate the body's resistance," modern clinical applications of EA combined with specific acupoint regimens (e.g., ST36, Sanyinjiao) have effectively alleviated cancer-related pain, chemotherapy-induced side effects, and fatigue. This study will evaluate the safety and immunosensitization effects of ST36 EA combined with PD-1 inhibitors in non-small cell lung cancer patients, employing 1 mA electroacupuncture for 3 consecutive days to activate immune responses. By leveraging acupuncture-induced immune remodeling, this approach aims to provide a novel integrative medicine strategy to overcome resistance to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 years at the time of written informed consent, of either sex;
2. Histologically or cytologically confirmed diagnosis of extensive-stage small cell lung cancer (SCLC) or non-small cell lung cancer (NSCLC) receiving neoadjuvant immunotherapy;
3. Undergoing standard first-line treatment with chemotherapy plus immunotherapy
4. ECOG performance status score of 0-2;
5. Life expectancy >3 months;
6. At least one measurable target lesion per RECIST 1.1 criteria:
7. Tumor lesions with a long axis ≥10 mm on CT scan (slice thickness ≤5 mm);
8. Lymph node lesions with a short axis ≥10 mm on CT scan;
9. Previously irradiated or locally treated lesions may be designated as target lesions if documented tumor progression post-treatment.
10. Adequate major organ function within 14 days prior to randomization, defined by the following laboratory parameters without blood transfusions, growth factors, albumin, or blood products:
11. Hematological tests: Hemoglobin ≥80 g/L; Absolute neutrophil count >1.5×10⁹/L; Platelet count ≥90×10⁹/L;
12. Biochemical tests: Total bilirubin ≤1.5×ULN (upper limit of normal); ALT/AST ≤2.5×ULN; Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min (Cockcroft-Gault formula);
13. Coagulation tests: Prothrombin time (PT) and INR ≤1.5×ULN (unless on warfarin anticoagulation);
14. Cardiac evaluation: Left ventricular ejection fraction (LVEF) ≥50% by Doppler echocardiography.
15. Voluntary participation with signed informed consent, good compliance, and willingness of the patient and their family to cooperate with survival follow-up.

Exclusion Criteria:

1. Pregnant participants;
2. Post-organ transplant patients;
3. Patients with uncontrolled diabetes mellitus, severe cardiac, central nervous system, psychiatric disorders, or coagulopathy;
4. Patients with severe malnutrition;
5. Patients with implanted cardiac pacemakers;
6. Patients with bleeding disorders;
7. Patients with a history of severe allergies or anaphylaxis;
8. Patients with skin infections, lesions, ulcers, or scars at the ST36 (Zusanli) acupoint site;
9. Patients with metal allergy, severe needle phobia, or intolerance to electroacupuncture therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Neoadjuvant Immunotherapy Conversion Rate | Baseline, After neoadjuvant immunotherapy (2-3 cycle, about 2 months after baseline)

SECONDARY OUTCOMES:
Peripheral blood immune cell alterations | Baseline (Day 1), end of Cycle 1 (21 days), Cycle 2 (42 days), and Cycle 3 (63 days). Each immunotherapy cycle is 21 days
  Peripheral blood immune cell alterations assessed by flow cytometry: CD4+/CD8+ T-cell ratio, Tregs, and NK cell subsets
Serum and Urine dopamine pathway and metabolites | Baseline (Day 1), end of Cycle 1 (21 days), Cycle 2 (42 days), and Cycle 3 (63 days). Each immunotherapy cycle is 21 days
  Serum norepinephrine and epinephrine concentrations analyzed via mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Xuelei Ma, MD, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol